CLINICAL TRIAL: NCT06726785
Title: Gene Expression Changes on Extended Use of Dopamine Agonists in Restless Legs Syndrome (RLS)
Brief Title: Observe Change in Nasal Swab DRD2 Gene Expression in Restless Legs Syndrome (RLS) Patients on Prolonged Dopamine Agonist Treatment
Acronym: RLS-DRD2gene
Status: Recruiting | Type: Observational
Sponsor: HBC Immunology Inc (Industry)
Responsible Party: Principal Investigator, Bomi Framroze, Principal Investigator, HBC Immunology Inc
Other Study IDs: RLS_IRB_12415
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Restless Leg Syndrome (RLS)
Keywords: restless leg syndrome; RLS; neurological
MeSH Terms: conditions — Restless Legs Syndrome; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary Endpoint: Nasal epithelial cell analysis for changes in dopaminergic genes expression between the two groups .
  Secondary Endpoints: Exploratory nasal epithelial cell swab data analysis for changes in other neural pathway genes expression between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study aims to observe changes in dopaminergic genes expression in peripheral tissue upon prolonged dopamine agonist treatment on patients with Restless Legs Syndrome (RLS). Similar studies in Parkinson's disease have shown changes in alpha-synuclein expression, which might offer insights into the dopaminergic gene regulation seen in RLS. The dopamine agonist drugs to be included in this study are: Pramipexole (Mirapex), Ropinirole (Requip), Rotigotine (Neupro), Apomorphine (Apokyn), Bromocriptine (Parlodel). Specifically, the study will collect nasal swabs of participants partitioned into two groups, those who have not used a dopamine agonist or been on a dopamine agonist for less than 1 month compared to those who have been on the medication for 6 or more months. This research could provide insight into changes in dopaminergic gene expression associated with Augmentation Syndrome (AS) which occurs after long term dopamine agonist treatment in RLS patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide Informed Consent
* Clinical diagnosis of Restless Legs Syndrome (RLS)
* On-going Treatment with a dopamine agonist

Exclusion Criteria:

* Use of any medication that might affect nasal epithelial cell collection with a nasal swab

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Diagnosed with RLS and on Dopamine Agonist treatments.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
To analyze the effect of duration of dopamine agonist treatments for changes in dopaminergic genes expression using nasal epithelial cells. | 1 week
  Gene expression will be measured and reported as the Fold change, which is the ratio of expression levels between the DRD2 experimental gene vs GAPDH housekeeping gene expression and reported as the Fold change which will indicate the magnitude of upregulation or downregulation of the DRD2 gene. A fold change >= 2 will be used as the minimum baseline to indicate upregulation and a fold change < = 1/2 will be used as the minimum baseline to indicate downregulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Alethios Inc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No